CLINICAL TRIAL: NCT05630950
Title: Low-dose CT Screening for Lung Cancer Combined to Different Smoking Cessation Methods in Finland
Brief Title: LDCT-SC-FI Low-dose CT Screening for Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Koivunen, MD PhD, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EETTKM 21/2022
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation application (Experimental)
  Interventions: Device: Smoking cessation mobile application
- Written smoking cessation information (Active Comparator)
  Interventions: Behavioral: Written material for smoking cessation

INTERVENTIONS:
Device: Smoking cessation mobile application — Mobile application for smoking cessation.
  Arms: Smoking cessation application
Behavioral: Written material for smoking cessation — Written material for smoking cessation
  Arms: Written smoking cessation information

SUMMARY:
This is a randomized phase II trial investigating different smoking cessation methods in study subjects undergoing lung cancer screening with low-dose CT (LDCT). The study also evaluates feasibility and outcomes of LDCT screening and potential biomarkers and AI-based evaluation on CT-scans. The study subjects fulfilling I/E-criteria are randomized in 1:1 fashion to yearly LDCT for two rounds with standard smoking cessation (control) or same LDCT approach combined to mobile application based smoking cessation (intervention).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Age between 50-74
* Smoked ≥ 15 cigarettes/day for ≥ 25 years or smoked ≥ 10 cigarettes/day for ≥ 30 years and are active smokers (smoking during the last two weeks)
* Access to a smartphone (iPhone or Android)

Exclusion Criteria:

* A moderate or bad self-reported health; e.g. unable to climb two flights of stairs
* Body weight ≥ 140 kilogram
* Current or past melanoma, lung, renal or breast cancer
* A chest CT examination less than one year before inclusion
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Subject is unwilling or unable to comply with treatment and trial instructions
* Any condition that study investigators consider an impediment to safe trial participation

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of active smokers at 3 months | 3 months
  The percentage of subjects who are actively smoking at 3 months after inclusion between the study arms

SECONDARY OUTCOMES:
Number of subjects who have reduced the amount of smoked cigrattes/d at 3 months | 3 months
  The percentage of subjects who have reduced the amount of smoked cigrattes/d at 3 months after inclusion compared to between the study arms
Number of subjects who have reduced the amount of smoked cigrattes/d at 6 months | 6 months
  The percentage of subjects who have reduced the amount of smoked cigrattes/d at 6 months after inclusion compared to baseline between the study arms
The reduction in number of smoked cigarettes/d at 3 months | 3 months
  Magnitude of reduction in number of cigarettes consumed/d at 3 month after inclusion compared to baseline between the study arms.
The reduction in number of smoked cigarettes/d at 6 months | 6 months
  Magnitude of reduction in number of cigarettes consumed/d at 6 month after inclusion compared to baseline between the study arms.
The percentage of reduction in number of smoked cigarettes/d at 3 months | 3 months
  Percentage of reduction in number of cigarettes consumed/d at 3 month after inclusion compared to baseline between the study arms.
The percentage of reduction in number of smoked cigarettes/d at 6 months | 6 months
  Percentage of reduction in number of cigarettes consumed/d at 6 month after inclusion compared to baseline between the study arms.
Sensitivity of CT screening in the whole cohort | At 2 years
  The amount of true positive CT scans for lung cancer compared to false negative CT scans for lung cancer.
Costs related to CT screening including additional investigations | At 2 years
  The cumulative cost of diagnostic investigations per study subject.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Oulu University Hospital, Oulu
  - Vaasa Central Hospital, Vaasa

IPD SHARING:
Plan to Share IPD: No
National legislation does not make it possible to share clinical data.

REFERENCES:
- [Derived] Iivanainen S, Kurtti A, Wichmann V, Andersen H, Jekunen A, Kaarteenaho R, Vasankari T, Koivunen JP. Smartphone application versus written material for smoking reduction and cessation in individuals undergoing low-dose computed tomography (LDCT) screening for lung cancer: a phase II open-label randomised controlled trial. Lancet Reg Health Eur. 2024 May 25;42:100946. doi: 10.1016/j.lanepe.2024.100946. eCollection 2024 Jul. PMID 39070744